CLINICAL TRIAL: NCT00411749
Title: V501 Phase II Immunogenicity Study in Females Aged 9 to 17 Years
Brief Title: V501 Immunogenicity Study in Females Age 9 to 17 Years (V501-028)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-028; 2006_052
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- V501 (Experimental): V501 vaccination Quadrivalent HPV (Types 6, 11, 16,
  18) L1 VLP Vaccine Injection
  cervix cancer exgenlesion Vaccination at Day 1, Month 2, and Month 6. Total 3 vaccinations. 0.5 mL intramuscular dose of V501 (HPV L1 Virus-Like Particle [VLP] Type 6,
  Type 11, Type 16, Type 18) or placebo at Day 1, Month 2 and Month 6.
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (V501)
- Placebo (Placebo Comparator): Placebo vaccination, Placebo 0.5 ml injection in 3 dosing regimen
  Interventions: Biological: Comparator: Placebo (unspecified)

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (V501) — V501; Gardasil, 0.5 ml injection in 3 dosing regimen
  Other Names: V501; Gardasil
  Arms: V501
Biological: Comparator: Placebo (unspecified) — Placebo 0.5 ml injection in 3 dosing regimen
  Arms: Placebo

SUMMARY:
The study evaluates the immunogenicity, safety and tolerability of V501 in preadolescent females

ELIGIBILITY:
Inclusion Criteria:

* Virginal Female Subject Aged 9 To 17 Years

Exclusion Criteria:

* Male Subject

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2006-12-11 (Actual); Primary Completion 2009-09-18 (Actual); Study Completion 2009-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Murata S, Shirakawa M, Sugawara Y, Shuto M, Sawata M, Tanaka Y. Post-hoc analysis of injection-site reactions following vaccination with quadrivalent human papillomavirus vaccine in Japanese female clinical trial participants. Papillomavirus Res. 2020 Dec;10:100205. doi: 10.1016/j.pvr.2020.100205. Epub 2020 Aug 19. PMID 32827835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 8 sites in Japan from 2006 to 2009.
Groups:
- V501: V501 vaccination: Gardasil, 0.5 ml injection in 3 dosing regimen. Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (V501)
- Placebo: Placebo vaccination 0.5 ml injection in 3 dosing regimen.
Period: Overall Study
Arm/Group | V501 | Placebo
Started | 82 | 25
Vaccinated | 82 | 25
Completed | 82 (Completed at 24 month after vaccination series (Month 30). Subjects were followed until Month 30) | 25 (Completed at 1 month after vaccination series (Month 7). Subjects were followed until Month 7)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V501 | Placebo | Total
Number analyzed (Participants) | 82 | 25 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (2.4) | 12.6 (2.6) | 12.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 25 | 107
  Male | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kilogram] | 45.5 (10.8) | 45.2 (9.6) | 45.4 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Human Papilloma Virus (HPV) 6 Serum Antibody Titer at One Month After Completed Vaccination Series
Description: Month 7 HPV Competitive Luminex immunoassay (cLIA) Geometric Mean Titers (GMT) by vaccine group.
  The limit of detection of the assay was 7 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "7.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: The per protocol immunogenicity population includes all subjects who were not general protocol violators, received all 3 vaccinations within acceptable day ranges, were seronegative at Day 1 for the relevant HPV type, and a Month 7 serum sample collected within an acceptable time range.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers (mMU/mL)
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 80 | 25
Geometric Mean Titers (mMU/mL) | 674.5 [528.6 to 860.8] | 7.0 [7.0 to 8.4]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Human Papilloma Virus (HPV) 11 Serum Antibody Titer at One Month After Completed Vaccination Series
Description: Month 7 HPV Competitive Luminex immunoassay (cLIA) Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 8 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "8.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers (mMU/mL)
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 80 | 25
Geometric Mean Titers (mMU/mL) | 944.5 [755.3 to 1181.0] | 8.0 [8.0 to 8.5]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Human Papilloma Virus (HPV) 16 Serum Antibody Titer at One Month After Completed Vaccination Series
Description: Month 7 HPV Competitive Luminex immunoassay (cLIA) Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 11 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "11.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers (mMU/mL)
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 82 | 25
Geometric Mean Titers (mMU/mL) | 4275.4 [3375.4 to 5415.4] | 11.0 [11.0 to 13.5]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Human Papilloma Virus (HPV) 18 Serum Antibody Titer at One Month After Completed Vaccination Series
Description: Month 7 HPV Competitive Luminex immunoassay (cLIA) Geometric Mean Titers by vaccine group.
  The limit of detection of the assay was 10 mMU/ml. GMTs and confidence limits below the limit of detection are shown as "10.0".
Time Frame: At one month after completed vaccination series (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers (mMU/mL)
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 82 | 25
Geometric Mean Titers (mMU/mL) | 829.2 [642.3 to 1070.5] | 10.0 [10.0 to 10.1]
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: HPV 6, 11, 16 and 18 Serum Antibody Titer at 24 Month After Completed Vaccination Series
Description: Month 30 HPV cLIA Geometric Mean Titers by vaccine group.
Time Frame: 24 month after completed vaccination series (Month 30)
Population: The per protocol immunogenicity population includes all subjects who were not general protocol violators, received all 3 vaccinations within acceptable day ranges, were seronegative at Day 1 for the relevant HPV type, and a Month 30 serum sample collected within an acceptable time range.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers (mMU/mL)
Groups:
- V501-HPV 6: HPV 6 serum antibody titer measured in V501 vaccination group
- V501-HPV 11: HPV 11 serum antibody titer measured in V501 vaccination group
- V501-HPV 16: HPV 16 serum antibody titer measured in V501 vaccination group
- V501-HPV 18: HPV 18 serum antibody titer measured in V501 vaccination group
Arm/Group | V501-HPV 6 | V501-HPV 11 | V501-HPV 16 | V501-HPV 18
Number analyzed (Participants) | 79 | 80 | 82 | 82
Geometric Mean Titers (mMU/mL) | 155.2 [126.2 to 190.9] | 198.2 [160.9 to 244.2] | 617.1 [491.7 to 774.5] | 90.0 [68.8 to 117.8]
Statistical Analysis 1: Comparison: V501-HPV 6; Test type: Superiority or Other; Geometric Mean = 155.2, 95% CI 2-sided [126.2 to 190.9]
Statistical Analysis 2: Comparison: V501-HPV 11; Test type: Superiority or Other; Geometric Mean = 198.2, 95% CI 2-sided [160.9 to 244.2]
Statistical Analysis 3: Comparison: V501-HPV 16; Test type: Superiority or Other; Geometric Mean = 617.1, 95% CI 2-sided [491.7 to 774.5]
Statistical Analysis 4: Comparison: V501-HPV 18; Test type: Superiority or Other; Geometric Mean = 90.0, 95% CI 2-sided [68.8 to 117.8]

ADVERSE EVENTS:
Time Frame: Serious Adverse Event (SAE) data were collected from the entire period of the study. Other non serious AE data were collected from Day 1 to Day 15 following vaccination.
Description: All adverse events described in case report forms were tabulated by converting them to the preferred term (PT) and classifying them by primary system organ class (PSOC) using the International Conference on Harmonisation (ICH) medical dictionary for regulatory activities (MedDRA) Ver. 9.0.
Arm/Group | V501 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/82 | 0/25
Other Adverse Events (participants affected / at risk) | 77/82 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V501 (N=82) | Placebo (N=25)
Strabismus congenital (Congenital, familial and genetic disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V501 (N=82) | Placebo (N=25)
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Injection site erythema (General disorders) | 35 | 5
Injection site haemorrhage (General disorders) | 0 | 1
Injection site pain (General disorders) | 69 | 19
Injection site pruritus (General disorders) | 12 | 1
Malais (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 1
Injection site swelling (General disorders) | 38 | 4
Injection site discomfort (General disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 9 | 5
Platelet count increased (Investigations) | 3 | 0
Protein urine present (Investigations) | 4 | 2
Headache (Nervous system disorders) | 9 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.